CLINICAL TRIAL: NCT02389621
Title: A Phase 3 Randomised, Double-blind, Placebo-controlled Study to Assess the Safety and Efficacy of S-888711 (Lusutrombopag) for the Treatment of Thrombocytopenia in Patients With Chronic Liver Disease Undergoing Elective Invasive Procedures (L-PLUS 2)
Brief Title: Safety and Efficacy Study of Lusutrombopag for Thrombocytopenia in Patients With Chronic Liver Disease Undergoing Elective Invasive Procedures
Acronym: L-PLUS 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1423M0634; 2014-004942-91 (EudraCT Number: European Commission)
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Chronic Liver Disease; Thrombocytopenia
Keywords: Elective invasive procedures
MeSH Terms: conditions — Thrombocytopenia | interventions — lusutrombopag

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lusutrombopag (Experimental): Lusutrombopag 3 mg once daily for up to 7 days.
  Interventions: Drug: Lusutrombopag
- Placebo (Placebo Comparator): Placebo once daily for up to 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lusutrombopag — Tablets for oral administration
  Other Names: S-888711
  Arms: Lusutrombopag
Drug: Placebo — Tablets for oral administration
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to compare the efficacy of lusutrombopag with placebo for the treatment of thrombocytopenia in patients with chronic liver disease who are undergoing elective invasive procedures.

DETAILED DESCRIPTION:
The study consists of 3 periods: a screening period (up to 28 days prior to randomization), a treatment period of 7 days (Days 1 to 7 during which study drug is to be administered for 4 to 7 days), and a posttreatment period (through 28 days posttreatment).

Once-daily treatment with lusutrombopag 3 mg or placebo is to commence on Day 1 and continue for up to 7 days. Platelet count is to be determined on Days 5, 6, and 7 prior to administration of study drug; if a participant meets the administration stopping criterion (ie, platelet count ≥ 50 × 10⁹/L with an increase of ≥ 20 × 10⁹/L from baseline), no additional dose of study drug is to be administered. The planned invasive procedure is to be performed in the posttreatment period between Days 9 and 14. Platelet count for determination of the need for platelet transfusion is to be determined on or after Day 8, but no more than 2 days prior to the invasive procedure; a platelet transfusion is required if the platelet count is < 50 × 10⁹/L.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the study and comply with all study procedures.
2. Willing to provide written informed consent prior to Screening.
3. Male or female.
4. 18 years of age or older at the time of signing informed consent.
5. Platelet count < 50 × 10^9/L at baseline on Day 1 prior to randomization.
6. Undergoing an elective invasive procedure.
7. In the opinion of the investigator, able to meet study requirements.
8. Male patients who are sterile or who agree to use an appropriate method of contraception (including use of a condom with spermicide) from Screening to completion of the Post-treatment Period.
9. Female patients who are not postmenopausal or surgically sterile need to agree to use a highly effective contraception (including contraceptive implant, injectable contraceptive, combination hormonal contraceptive [including vaginal rings], intrauterine contraceptive device or vasectomised partner) from Screening to completion of the Post-treatment Period. Barrier method with or without spermicide, double barrier contraception and oral contraceptive pill are insufficient methods on their own.

Exclusion Criteria:

1. Any of the following diseases:

   * hematopoietic tumor
   * aplastic anemia
   * myelodysplastic syndrome
   * myelofibrosis
   * congenital thrombocytopenia
   * drug-induced thrombocytopenia
   * generalized infection requiring treatment except for viral liver disease
   * immune thrombocytopenia.
2. History of splenectomy.
3. History of liver transplantation.
4. Any of the following at Screening:

   * hepatic encephalopathy uncontrolled by drugs
   * ascites uncontrolled by drugs.
5. Portal vein tumor embolism.
6. Known to be positive for the human immunodeficiency virus.
7. Past or present thrombosis or prothrombotic condition (e.g., cerebral infarction, myocardial infarction, angina pectoris, coronary artery stent placement, angioplasty, coronary artery bypass grafting, congestive heart failure [New York Heart Association Grade III/IV], arrhythmia known to increase the risk of thromboembolic events [atrial fibrillation], pulmonary thromboembolism, deep vein thrombosis, or disseminated intravascular coagulation syndrome).
8. History or evidence of any of the following diseases:

   * congenital thrombotic disease (eg, antithrombin deficiency, protein C deficiency, protein S deficiency, or coagulation factor [Factor V Leiden] mutation)
   * acquired thrombotic disease (eg, antiphospholipid antibody syndrome, paroxysmal nocturnal hemoglobinuria, hyperhomocysteinemia, or increased factor VIII)
   * Budd Chiari syndrome.
9. Portal vein thrombosis based on ultrasound, computed tomography (CT), or magnetic resonance imaging (MRI) within 28 days prior to randomization or a history of portal vein thrombosis.
10. Absence of hepatopetal blood flow in the main trunk of the portal vein as demonstrated by Doppler ultrasonography within 28 days prior to randomization.
11. History or evidence of disease associated with a risk of bleeding (e.g., coagulation factor deficiency or von Willebrand factor deficiency).
12. Bleeding score at randomization ≥ Grade 2 according to the World Health Organization (WHO) Bleeding Scale.
13. Any of the following drugs or therapies within 90 days prior to randomization:

    * anticancer drugs
    * interferon preparations
    * radiation therapy
    * exsanguination
    * other thrombopoietin receptor agonist
    * any investigational agent.
14. Any invasive procedure within 14 days prior to randomization.
15. Blood transfusion within 14 days prior to randomization.
16. Prior treatment with lusutrombopag (S-888711).
17. Pregnancy or lactation.
18. Known or suspected ongoing, active alcohol or substance abuse. Patients with a recent history who the investigator feels are able to comply with the study procedures and medications will be allowed to participate.
19. Considered ineligible by the investigator for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi

REFERENCES:
- [Derived] Flamm SL, Peck-Radosavljevic M, Fukuhara T, Bentley R, Katsube T, Ochiai T, Kano T, Tsukimura E, Sasaki R, Osaki Y. Pharmacokinetic Assessment and Treatment Effect of Lusutrombopag in Child-Pugh Class C Patients: Review of Patient Data from Two Clinical Studies and Post-Marketing Surveillance. Adv Ther. 2022 Sep;39(9):4285-4298. doi: 10.1007/s12325-022-02237-8. Epub 2022 Jul 29. PMID 35904722
- [Derived] Alkhouri N, Imawari M, Izumi N, Osaki Y, Ochiai T, Kano T, Bentley R, Trevisani F. Lusutrombopag Is Safe and Efficacious for Treatment of Thrombocytopenia in Patients With and Without Hepatocellular Carcinoma. Clin Gastroenterol Hepatol. 2020 Oct;18(11):2600-2608.e1. doi: 10.1016/j.cgh.2020.03.032. Epub 2020 Mar 20. PMID 32205226

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 138 sites in 22 countries (Argentina, Australia, Austria, Belgium, Canada, Czech Republic, France, Germany, Hungary, Israel, Italy, Poland, Republic of Korea, Romania, Russian Federation, Spain, Taiwan, Thailand, Turkey, Ukraine, United Kingdom, and United States of America).
Pre-assignment Details: The study consisted of a screening period (up to 28 days), a treatment period of 7 days, and a posttreatment period (through 28 days posttreatment).
  Randomization was stratified by the primary invasive procedure (ie, liver ablation/coagulation or other invasive procedures) and baseline platelet count (< 35 × 10⁹/L or ≥ 35 × 10⁹/L).
Period: Treatment Period
Arm/Group | Lusutrombopag | Placebo
Started | 108 | 107
Received Study Drug | 107 | 107
Completed | 107 | 106
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Posttreatment Period
Arm/Group | Lusutrombopag | Placebo
Started | 107 | 106
Completed | 98 | 102
Not Completed | 9 | 4
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Other - Miscellaneous | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lusutrombopag | Placebo | Total
Number analyzed (Participants) | 108 | 107 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (11.6) | 56.1 (11.0) | 55.7 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 38 | 81
  Male | 65 | 69 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 12 | 26
  Not Hispanic or Latino | 93 | 95 | 188
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 15 | 17 | 32
  Black or African American | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 85 | 86 | 171
  Other | 3 | 0 | 3
  Not provided | 2 | 4 | 6
Planned Invasive Procedure [Count of Participants; unit: Participants]
  Liver ablation/ coagulation | 7 | 5 | 12
  Other | 101 | 102 | 203
Baseline Platelet Count [Count of Participants; unit: Participants]
  < 35 × 10⁹/L | 36 | 38 | 74
  ≥ 35 × 10⁹/L | 71 | 68 | 139
  Missing | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Required No Platelet Transfusion Prior to the Primary Invasive Procedure and No Rescue Therapy For Bleeding From Randomization Through 7 Days After the Primary Elective Procedure
Description: Participants were considered as meeting the primary endpoint if all of the following conditions were satisfied:
  * Required no platelet transfusion from the date of randomization through at least 7 days after the primary invasive procedure
  * Did not receive the following rescue therapy for bleeding from the date of randomization through 7 days after the primary invasive procedure
    * Platelet preparations
    * Other blood preparations, including red blood cells and plasma
    * Volume expanders
  * Underwent an invasive procedure. Participants who received at least one platelet transfusion prior to the primary invasive procedure, received at least one rescue therapy for bleeding from the date of randomization through 7 days after the primary invasive procedure, discontinued from the study before undergoing the primary invasive procedure, or did not undergo an invasive procedure were considered as not meeting the primary endpoint.
Time Frame: From Randomization to 7 days after the invasive procedure, up to approximately 21 days.
Population: All randomized participants (intent-to-treat population)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lusutrombopag | Placebo
Number analyzed (Participants) | 108 | 107
percentage of participants | 64.8 [55.0 to 73.8] | 29.0 [20.6 to 38.5]
Statistical Analysis 1: Comparison: Lusutrombopag vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Statistical tests were performed at a 2-sided significance level of 0.05; Adjusted using the stratification factors of platelet count at randomization and the planned primary invasive procedure; Difference = 36.7, 95% CI 2-sided [24.9 to 48.5]

2. Secondary Outcome: Percentage of Participants Who Required no Platelet Transfusion During the Study
Description: Participants who did not undergo the invasive procedure were considered as having received platelet transfusion.
Time Frame: From Day 1 to end of the posttreatment period, 35 days.
Population: All randomized participants (intent-to-treat population)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lusutrombopag | Placebo
Number analyzed (Participants) | 108 | 107
percentage of participants | 63.0 [53.1 to 72.1] | 29.0 [20.6 to 38.5]
Statistical Analysis 1: Comparison: Lusutrombopag vs Placebo; Test type: Superiority — A gatekeeping procedure was employed for sequentially testing the prespecified important secondary endpoints, identified as the most clinically relevant endpoints. If the primary endpoint was statistically significant, the secondary endpoints were tested at the 0.05 level (2-sided) in sequence; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted for the stratification factors of platelet count at randomization and the planned primary invasive procedure; Difference = 34.8, 95% CI 2-sided [22.8 to 46.8]

3. Secondary Outcome: Percentage of Participants With a Response
Description: A response was defined as a platelet count of ≥ 50 × 10⁹/L with an increase of ≥ 20 × 10⁹/L from Baseline at any time during the study. Participants who met this response criterion only after platelet transfusion were considered as nonresponders.
Time Frame: From Day 1 to the end of the posttreatment period, 35 days.
Population: All randomized participants (intent-to-treat population)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lusutrombopag | Placebo
Number analyzed (Participants) | 108 | 107
percentage of participants | 64.8 [55.0 to 73.8] | 13.1 [7.3 to 21.0]
Statistical Analysis 1: Comparison: Lusutrombopag vs Placebo; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted for the stratification factors of platelet count at randomization and the planned primary invasive procedure; Difference = 52.5, 95% CI 2-sided [42.0 to 62.9]

4. Secondary Outcome: Duration of Increase in Platelet Count to ≥ 50 × 10⁹/L
Description: The duration of the increase in platelet count was defined as the number of days during which the platelet count was maintained as ≥ 50 × 10⁹/L.
Time Frame: From Day 1 to the end of the posttreatment period, 35 days.
Population: All randomized participants with available data
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Lusutrombopag | Placebo
Number analyzed (Participants) | 107 | 107
days | 15.11 [6.59 to 23.88] | 0.98 [0.00 to 9.22]
Statistical Analysis 1: Comparison: Lusutrombopag vs Placebo; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0002, van Elteren test; van Elteren test stratified by platelet transfusion during the study

5. Secondary Outcome: Duration of Increase in Platelet Count to ≥ 50 × 10⁹/L by Platelet Transfusion Status
Description: as for outcome 4
Time Frame: From Day 1 to the end of the posttreatment period, 35 days.
Population: All randomized participants with available data
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Lusutrombopag With Platelet Transfusion: Lusutrombopag 3 mg once daily for up to 7 days in participants who received platelet transfusion.
- Lusutrombopag Without Platelet Transfusion: Lusutrombopag 3 mg once daily for up to 7 days in participants who did not receive platelet transfusion.
- Placebo With Platelet Transfusion: Placebo once daily for up to 7 days in participants who received platelet transfusion.
- Placebo Without Platelet Transfusion: Placebo once daily for up to 7 days in participants who did not receive platelet transfusion.
Arm/Group | Lusutrombopag With Platelet Transfusion | Lusutrombopag Without Platelet Transfusion | Placebo With Platelet Transfusion | Placebo Without Platelet Transfusion
Number analyzed (Participants) | 34 | 73 | 73 | 34
days | 1.73 [0.00 to 14.00] | 19.21 [12.64 to 28.00] | 0.00 [0.00 to 5.04] | 8.86 [0.00 to 18.73]
Statistical Analysis 1: Comparison: Lusutrombopag Without Platelet Transfusion vs Placebo With Platelet Transfusion; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, Wilcoxon rank sum test

6. Secondary Outcome: Percentage of Participants Who Required Rescue Therapy for Bleeding During the Study
Description: Participants who received rescue therapy for bleeding events during the study. Platelet preparations, other blood preparations (including red blood cells and plasma), and volume expanders were considered as rescue therapy for bleeding events.
Time Frame: From Day 1 to the end of the possttreatment period, 35 days.
Population: All randomized participants (intent-to-treat population)
Measure: Number; unit: percentage of participants
Arm/Group | Lusutrombopag | Placebo
Number analyzed (Participants) | 108 | 107
percentage of participants | 0.0 | 1.9

7. Secondary Outcome: Number of Participants With Specified Total Number of Platelet Transfusions
Description: The number of transfusions administered to each patient were collected over the duration of the trial. The data are presented as the number of patients with the highest total number of transfusions followed by the next highest number of transfusions, etc.
Time Frame: From Day 1 to the end of the posttreatment period, 35 days.
Population: All randomized participants (intent-to-treat population)
Measure: Count of Participants; unit: Participants
Arm/Group | Lusutrombopag | Placebo
Number analyzed (Participants) | 108 | 107
Participants
  No transfusions | 74 | 34
  One transfusion | 34 | 61
  Two transfusions | 0 | 6
  Three transfusions | 0 | 5
  Four transfusions | 0 | 0
  Five transfusions | 0 | 1

8. Secondary Outcome: Change From Baseline in Platelet Count Over Time
Time Frame: Baseline and Days 5, 6, 7, 8, 10, 12, 14, 17, 21, 28, and 35.
Population: All randomized participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: * 10⁹/L
Arm/Group | Lusutrombopag With Platelet Transfusion | Lusutrombopag Without Platelet Transfusion | Placebo With Platelet Transfusion | Placebo Without Platelet Transfusion
Number analyzed (Participants) | 34 | 74 | 73 | 34
* 10⁹/L
  Day 5: number analyzed (Participants) | 34 | 72 | 73 | 33
  Day 5 | 1.1 (6.5) | 10.4 (12.5) | 0.4 (6.6) | 6.1 (11.8)
  Day 6: number analyzed (Participants) | 34 | 70 | 73 | 31
  Day 6 | 5.1 (8.1) | 13.6 (15.7) | -0.6 (7.0) | 6.7 (12.4)
  Day 7: number analyzed (Participants) | 34 | 69 | 72 | 31
  Day 7 | 4.7 (7.9) | 20.6 (16.8) | 0.0 (7.7) | 6.7 (12.9)
  Day 8: number analyzed (Participants) | 31 | 69 | 68 | 32
  Day 8 | 7.7 (9.5) | 27.4 (21.5) | -0.1 (5.2) | 7.3 (13.5)
  Day 10: number analyzed (Participants) | 32 | 64 | 64 | 26
  Day 10 | 12.6 (10.6) | 36.7 (24.1) | 2.1 (11.0) | 12.7 (20.6)
  Day 12: number analyzed (Participants) | 27 | 63 | 70 | 26
  Day 12 | 15.4 (12.3) | 37.0 (18.5) | 3.1 (9.5) | 14.8 (24.0)
  Day 14: number analyzed (Participants) | 33 | 62 | 67 | 28
  Day 14 | 17.3 (19.3) | 33.5 (19.9) | 4.0 (11.8) | 12.8 (28.1)
  Day 17: number analyzed (Participants) | 25 | 58 | 61 | 22
  Day 17 | 17.1 (23.4) | 27.2 (21.1) | 1.9 (9.0) | 17.0 (27.7)
  Day 21: number analyzed (Participants) | 32 | 67 | 66 | 29
  Day 21 | 9.8 (16.0) | 20.9 (20.3) | 2.5 (9.0) | 13.2 (20.7)
  Day 28: number analyzed (Participants) | 31 | 63 | 67 | 29
  Day 28 | 1.7 (11.4) | 12.4 (18.8) | 2.0 (8.9) | 10.1 (17.6)
  Day 35: number analyzed (Participants) | 32 | 64 | 69 | 31
  Day 35 | -1.3 (6.2) | 9.4 (19.3) | 0.7 (9.1) | 6.0 (15.9)

9. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Time Frame: From first dose of study drug to 28 days after the last dose, 35 days.
Population: All randomized participants who received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Lusutrombopag | Placebo
Number analyzed (Participants) | 107 | 107
Participants
  All adverse events | 51 | 52
  Serious adverse events | 7 | 7
  Adverse events with outcome of death | 3 | 0
  AEs leading to discontinuation of study drug | 0 | 1
  Treatment-related adverse events | 6 | 13

10. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Lusutrombopag
Time Frame: Day 5, predose and 2, 4, 6, 8, 24, and 48 hours post-dose (24 and 48 hours post-dose = Day 6 and Day 7 prior to dose on that day).
Population: Participants in the intensive pharmacokinetic (PK) sampling group with at least 1 PK parameter estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Lusutrombopag
Number analyzed (Participants) | 9
ng/mL | 157 (34.7)

11. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Lusutrombopag
Time Frame: as for outcome 10
Population: Participants in the intensive pharmacokinetic (PK) sampling group with at least 1 PK parameter estimated.
Measure: Median (Full Range); unit: hours
Arm/Group | Lusutrombopag
Number analyzed (Participants) | 9
hours | 5.95 [2.03 to 7.85]

12. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Dosing Interval τ (AUC0-τ) for Lusutrombopag
Time Frame: as for outcome 10
Population: Participants in the intensive pharmacokinetic (PK) sampling group with at least 1 PK parameter estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Lusutrombopag
Number analyzed (Participants) | 9
ng*hr/mL | 2737 (36.1)

13. Secondary Outcome: Apparent Total Clearance (CL/F) of Lusutrombopag
Time Frame: as for outcome 10
Population: Participants in the intensive pharmacokinetic (PK) sampling group with at least 1 PK parameter estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Lusutrombopag
Number analyzed (Participants) | 9
L/h | 1.10 (36.1)

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 28 days after last dose, 35 days
Arm/Group | Lusutrombopag | Placebo
All-Cause Mortality (participants affected / at risk) | 3/107 | 0/107
Serious Adverse Events (participants affected / at risk) | 7/107 | 7/107
Other Adverse Events (participants affected / at risk) | 23/107 | 22/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lusutrombopag (N=107) | Placebo (N=107)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Anemia (Blood and lymphatic system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 2
Encephalopathy (Nervous system disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Vessel perforation (Vascular disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Multiorgan failure (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lusutrombopag (N=107) | Placebo (N=107)
Nasopharyngitis (Infections and infestations) | 3 | 0
Headache (Nervous system disorders) | 6 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 5
Nausea (Gastrointestinal disorders) | 2 | 4
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3
Ascites (Gastrointestinal disorders) | 2 | 3
Diarrhea (Gastrointestinal disorders) | 3 | 2
Fatigue (General disorders) | 3 | 7
Edema peripheral (General disorders) | 3 | 4
Pyrexia (General disorders) | 3 | 2
Procedural pain (Injury, poisoning and procedural complications) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2015-02-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT02389621/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT02389621/SAP_001.pdf